CLINICAL TRIAL: NCT05521204
Title: A Study of Olverembatinib in the Treatment of Myeloid/Lymphoid Tumors With FGFR1 Rearrangement
Brief Title: Olverembatinib for FGFR1-rearranged Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-FGFR1
Record Dates: First submitted 2022-08-27; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Myeloproliferative Neoplasm; Acute Leukemia
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: Olverembatinib

INTERVENTIONS:
Drug: Olverembatinib — Given PO

SUMMARY:
FGFR1-rearranged myeloid/lymphoid neoplasms are a rare hematologic malignancy with very poor outcome despite intensive chemotherapy. The only curative option is thought to be allogeneic hematopoietic stem cell transplantation (HSCT) in remission.

This phase II study is aimed to evaluate the efficacy of Olverembatinib, consolidated with HSCT in the treatment of FGFR1-rearranged myeloid/lymphoid neoplasm.

DETAILED DESCRIPTION:
FGFR1-rearranged myeloid/lymphoid neoplasms are a rare and highly heterogeneous hematological malignancy, mainly manifested as myeloproliferative neoplasms (MPNs) or acute leukemia, including T cells or B cells Cell lymphoblastic leukemia/lymphoma (T-cell or B-cell-ALL/LBL), acute myeloid leukemia (AML) and mixed cell leukemia (MPAL).

To date, there is no standard treatment. Conventional chemotherapy is frequently ineffective. The only curative option is thought to be allogeneic HSCT at present, TKIs may offer a therapeutic alternative in patients not eligible for allogeneic HSCT or to bridge the time between diagnosis and allogeneic HSCT.

Third-generation TKIs Olverembatinib is a pan- FGFR1 kinase inhibitor, and is supposed to be effective to achieve bone marrow remission in FGFR1-rearranged myeloid/lymphoid neoplasms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed, progressed or relapsed myeloid/lymphoid neoplasms with FGFR1 rearrangement according to the WHO-2016 diagnostic criteria. Patients who have received allogeneic hematopoietic stem cell transplantation or ponatinib should be excluded.
2. ECOG score: MPNs patients, 0-3 points; AL patients, 0-2 points.
3. Expected survival period ≥12 weeks.
4. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Patients who have received allogeneic hematopoietic stem cell or ponatinib.
2. Human immunodeficiency virus (HIV) infection, or chronic infection with hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV positive).
3. Patients who are pregnant, planning to become pregnant or breastfeeding.
4. Patients who may not be able to complete all study visits or procedures required by the study protocol, including follow-up visits, and/or fail to comply with all required study procedures.
5. Patients who suffer from any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of the safety of the research drug.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Assessed at protocol-defined timepoints through end of study, up to approximately 48 months.
  The proportion of participants who achieve Overall Response (ORR) based on response criteria for myeloid/lymphoid neoplasms with FGFR1 rearrangement

SECONDARY OUTCOMES:
Event-free survival (PFS) | From the first day of treatment until any failure (resistant disease, relapse, or death), assessed up to 2 to 4 years.
  The Kaplan-Meier method will be used to assess EFS probabilities.
Overall survival (OS) | From the first day of treatment to time of death from any cause, assessed up 2 to 4 years.
  The Kaplan-Meier method will be used to assess OS probabilities.
Incidence of adverse events (AEs) | Up to approximately 2 to 4 years.
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The proportion of patients with AEs will be estimated, along with the Bayesian 95% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, Principal Investigator — First Affiliated Hospital of Soochow University
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China